CLINICAL TRIAL: NCT05266391
Title: Comparison of Clinical Results of Ultrasound-Guided Versus Blind Subacromial Corticosteroid Injections in Subacromial Impingement Syndrome
Brief Title: Injection Technique in Subacromial Impingement Syndrome
Acronym: SAIS
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: PMRTURKEY
Record Dates: First submitted 2022-02-28; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: patients who received US-guided subacromial corticosteroid injections
  Interventions: Other: subacromial corticosteroid injections
- group 2: patients who underwent blind subacromial corticosteroid injections
  Interventions: Other: subacromial corticosteroid injections

INTERVENTIONS:
Other: subacromial corticosteroid injections — Patients with SAIS whose application of corticosteroid in their injections were the same in terms of type and dose (1 ml betamethasone dipropionate + betamethasone sodium phosphate).

SUMMARY:
Since pain is usually accompanied by a substantial effect on daily life that results in the extensive use of healthcare resources. In subacromial impingement syndrome, shoulder pain affects the quality of life negatively by affecting upper extremity functions and interrupting night sleep. It is very important to control the pain in order to reduce the loss to the labor force and prevent the pain from becoming chronic. Various physical treatment methods such as ultrasound, hot pack, transcutaneous electrical nerve stimulation, etc., and injections or medical agents are recommended. This study aimed to compare the effects of ultrasound (US)-guided in comparison to landmark guided subacromial corticosteroids injection on shoulder range of motion (ROM), pain, and functional status in patients with subacromial impingement syndrome (SAIS).

DETAILED DESCRIPTION:
Patients were assigned to two groups: Group-1 included patients who received US-guided subacromial corticosteroid injections; Group-2 included patients who underwent blind subacromial corticosteroid injections. The primary Outcome Measure was a Visual analog scale. Secondary Outcome Measures were Shoulder joint range of motion (ROM), Shoulder Pain and Disability Index (SPADI), The Shortened Disabilities of the Arm, Shoulder and Hand Questionnaire (Quick DASH).

ELIGIBILITY:
Inclusion Criteria:

1. Shoulder posterolateral pain that increased with shoulder abduction,
2. Restriction of the shoulder passive and active range of motion (ROM),
3. Patients with positive Neer and Hawkins impingement test,
4. Patients with SAIS whose diagnosis was confirmed by magnetic resonance imaging (MRI), and
5. Patients with SAIS whose application of corticosteroid in their injections were the same in terms of type and dose (1 ml betamethasone dipropionate + betamethasone sodium phosphate).

Exclusion Criteria:

* Patients who received corticosteroid, local anesthetic, hyaluronic acid, and platelet-rich plasma injections in the shoulder in the last one year,
* patients who had previous history of surgery or fracture in their thorax, neck, upper extremity or shoulder joint,
* patients with a rheumatological, cognitive or psychiatric, central or peripheral neurological disease (stroke, spinal cord injury, brachial plexus injury, etc.),
* patients whose MRI presented a partial or complete rotator cuff tear, calcific tendinitis or labral tear.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of Subacromial impingement syndrome who underwent subacromial corticosteroid injections in our interventional physiatry clinic between September 2017 and February 2018 were included in this study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | Change from baseline visual analogue scale score at 1 month
  It is a scale scored from 0 to 10 to evaluate the severity of pain. Patients are asked to rate the pain they feel as '0' for no pain and '10' for the most severe pain they have encountered in their life

SECONDARY OUTCOMES:
Shoulder joint range of motion (ROM) | Change from baseline Shoulder joint range of motion at 1 month
  Shoulder ROMs were evaluated using a goniometer according to the standard method. Those with shoulder flexion lower than 160° and external rotation lower than 90° were recorded as restricted ROM
Shoulder Pain and Disability Index (SPADI) | Change from baseline Shoulder Pain and Disability Index at 1 month
  It is a scale in which pain and the limitation of shoulder function are evaluated between 0 and 10 points. Five items for the pain is scored 0 for "no pain," and 10 points for "most severe pain." Eight items for disability is scored 0 for "no difficulty," and 10 points for "difficulty requiring assistance." SPADI is a useful scale in both clinical practice and clinical trials, as it can also detect changes in the status of patients
The Shortened Disabilities of the Arm, Shoulder and Hand Questionnaire (Quick DASH) | Change from baseline The Shortened Disabilities of the Arm, Shoulder and Hand Questionnaire at 1 month
  It is used to evaluate the difficulty in performing various physical activities due to disabilities of the shoulder, arm or hand (6 items), the severity of pain and tingling (2 items), and the effect of the disability on social activities, work, and sleep (3 items). It is the shortened version of the DASH (Disabilities of the Arm, Shoulder and Hand Questionnaire) in 11 items. Each item is scored between 1 and 5. "No difficulty" is scored as 1 and "unable" is scored as 5 points. At least 10 of the 11 items must be answered. The final score is calculated from zero (no disability) to 100 (severe disability). Two optional items of the Quick DASH (work, and sports or music) were not used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye Ones, Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
results and conclusions